CLINICAL TRIAL: NCT03994367
Title: Animal and Plant Proteins and Glucose Metabolism
Acronym: HP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Bettina Mittendorfer, Senior Associate Dean for Research, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2097498
Record Dates: First submitted 2019-06-18; First posted 2019-06-21 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Metabolic Syndrome; Metabolic Syndrome, Protection Against; Glucose Metabolism Disorders
Keywords: High Protein; Metabolism; Diet
MeSH Terms: conditions — Metabolic Syndrome; Glucose Metabolism Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Standard protein (control) (No Intervention)
- High animal protein isolate (Experimental)
  Interventions: Other: High animal protein isolate
- High animal protein whole food (Experimental)
  Interventions: Other: High animal protein whole food
- High plant protein isolate (Experimental)
  Interventions: Other: High plant protein isolate
- High plant protein whole food (Experimental)
  Interventions: Other: High plant protein whole food

INTERVENTIONS:
Other: High animal protein isolate — Increased dietary protein content from animal protein isolates
  Arms: High animal protein isolate
Other: High animal protein whole food — Increased dietary protein content from animal protein whole food
  Arms: High animal protein whole food
Other: High plant protein isolate — Increased dietary protein content from plant protein isolates
  Arms: High plant protein isolate
Other: High plant protein whole food — Increased dietary protein content from animal protein whole food
  Arms: High plant protein whole food

SUMMARY:
The goal of this proposal is to determine the effect of a high protein diet in which the increase in protein intake is derived from different sources (animal vs plant and protein-rich whole foods vs protein isolates) on: i) liver and muscle insulin sensitivity; ii) the metabolic response to a meal, and iii) 24-h plasma concentration profiles of glucose, glucoregulatory hormones, and protein-derived metabolites purported to cause metabolic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* age: ≥21 and ≤70 years;
* BMI: >24.5 and <32.5 kg/m2;
* habitual protein intake <0.9 g/kg/day (assessed on 2 weekdays and 2 weekend days by using the HealthWatch 360 app); and
* weight stable (i.e., ≤3% change) and untrained (≤150 min of structured exercise/week) for at least 2 months before entering the study.

Exclusion Criteria:

* prediabetes or type 2 diabetes;
* evidence of chronic kidney disease by medical history or laboratory tests (glomerular filtration rate <60 ml/min/1.73 m2 or an albumin to creatinine ratio in urine ≥30 mg/g);
* vegetarians or vegans;
* intolerance or allergies to ingredients in the metabolic meal or intervention diet;
* take dietary supplements (e.g., pre- and probiotics, fiber, fish oil) or medications known to affect our study outcomes;
* received antibiotic or antifungal treatment (which affect the microbiome and therefore microbial metabolite production) 2 months before entering the study;
* consume tobacco products or excessive alcohol (women: >14 drinks/week; men: >21 drinks/week);
* evidence of significant organ system dysfunction or diseases (e.g., cirrhosis), and
* unwilling or unable to provide informed consent.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-07-12 (Actual); Primary Completion 2028-02-25 (Estimated); Study Completion 2028-04-25 (Estimated)

PRIMARY OUTCOMES:
24-hour plasma glucose concentration | up to 12 weeks after the intervention
Insulin sensitivity assessed as insulin-mediated glucose disposal during a hyperinsulinemic-euglycemic clamp procedure | up to 12 weeks after the intervention

SECONDARY OUTCOMES:
Postprandial plasma glucose concentration | up to 12 weeks after the intervention
mTOR signaling (phospho-S6 content) in circulating monocytes | up to 12 weeks after the intervention
Endothelial function, assessed as reactive hyperemia index | up to 12 weeks after the intervention
Postprandial plasma insulin concentration | up to 12 weeks after the intervention
Postprandial plasma amino acid concentration | up to 12 weeks after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Mittendorfer, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri School of Medicine, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No